CLINICAL TRIAL: NCT00003279
Title: The SILVA Study: Survival in an International Phase III Prospective Randomized LD Small Cell Lung Cancer Vaccination Study With Adjuvant BEC2 and BCG
Brief Title: Vaccination Therapy in Treating Patients With Limited-Stage Small Cell Lung Cancer
Acronym: SILVA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-08971; EORTC-08971; UCLA-9902001
Record Dates: First submitted 1999-11-01; First posted 2004-08-25 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — BCG Vaccine

INTERVENTIONS:
Biological: BCG vaccine
Biological: monoclonal antibody BEC2

SUMMARY:
RATIONALE: Vaccines may help the body build an immune response to kill tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of vaccination with monoclonal antibody BEC2 and BCG with that of no further therapy in treating patients who have limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the impact of adjuvant monoclonal antibody BEC2 and BCG on survival of patients with limited stage small cell lung cancer. II. Determine the safety of this regimen in these patients. III. Determine progression-free survival and quality of life of these patients treated with this regimen.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, Karnofsky performance status (60-70% vs 80-100%), and response to first-line combined modality treatment (complete vs partial). Within 3-7 weeks after completion of prior induction chemoradiotherapy, responding patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive best supportive care and are observed until disease progression is documented. Arm II: Patients receive adjuvant monoclonal antibody BEC2 and BCG intradermally on day 1 of weeks 0, 2, 4, 6, and 10. Treatment consists of 5 vaccinations over a period of 10 to 12 weeks in the absence of unacceptable toxicity or disease progression. Quality of life is assessed at baseline, at weeks 6, 12, and 24, and then every 6 months thereafter. Patients are followed every 3 months.

PROJECTED ACCRUAL: Approximately 500 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven limited stage small cell lung cancer (SCLC) Must have completed adequate first-line combined modality treatment comprising at least 4-6 courses of a 2-drug chemotherapy regimen and chest radiotherapy No evidence of disease progression or relapse Disease response (complete or partial) after treatment

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: WBC greater that 3,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: AST less than 1.5 times upper limit of normal Hepatitis B negative Renal: Not specified Cardiovascular: Adequate cardiac function Other: HIV negative Not pregnant or nursing Fertile patients must use effective contraception No prior malignancy within 5 years except adequately treated nonmelanomatous skin cancer or carcinoma in situ of the cervix No history of tuberculosis No grade 3 local skin toxicity reaction (ulceration) to 5 IU or greater of PPD test No active infections requiring systemic antibiotics, antiviral, or antifungal treatments No serious unstable chronic illnesses No psychological, familial, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior therapy with proteins of murine origin At least one month since prior immunotherapy No other concurrent immunotherapy Chemotherapy: See Disease Characteristics No concurrent chemotherapy Endocrine therapy: No concurrent chronic use of systemic corticosteroids Radiotherapy: See Disease Characteristics No concurrent radiotherapy including prophylactic cranial irradiation No prior spleen radiotherapy Surgery: No prior surgery for SCLC No prior splenectomy Other: No prior second-line therapy for SCLC At least one month since prior investigational agents No concurrent chronic use of systemic antihistamines or nonsteroidal anti-inflammatory drugs No concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 1998-03; Primary Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, MD, PhD, Study Chair — Free University Medical Center
Locations (77):
- United States (34):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Scripps Clinic and Research Foundation - La Jolla, La Jolla, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Colorado Permanente Medical Group, P.C., Denver, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Greenwich Hospital Association, Greenwich, Connecticut
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - Norwich Cancer Center, Norwich, Connecticut
  - Bennett Cancer Center, Stamford, Connecticut
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Memorial Regional Cancer Center, Hollywood, Florida
  - Mercy Hospital, Miami, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Columbia - HCA Cancer Research Network, North Miami Beach, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Georgia Cancer Specialists, Decatur, Georgia
  - Veterans Affairs Medical Center - West Roxbury, West Roxbury, Massachusetts
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Benefis Healthcare, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Southwest Cancer Clinic, Las Vegas, Nevada
  - University of Nevada - Reno, Reno, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Oklahoma Oncology Inc., Tulsa, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Charleston Area Medical Center, Charleston, West Virginia
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Australia (11):
  - Royal Prince Alfred Hospital, Sydney, Camperdown, New South Wales
  - Repatriation General Hospital, Concord, New South Wales
  - Newcastle Mater Misericordiae Hospital, Newcastle, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - NSW Breast Cancer Institute, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Center, East Bentweigh, Victoria
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Pulmologisches Zentrum Der Stadt Wien, Vienna (Wein), Austria
- U.Z. Gasthuisberg, Leuven, Belgium
- Germany (5):
  - Universitaetsklinikum Benjamin Franklin, Berlin
  - Asklepios Fachkliniken Munchen- Gauting, Gauting, Munich (Munchen)
  - Hospital Grosshansdorf, Großhansdorf
  - Thoraxklinik Rohrbach, Heidelberg
  - Marienhospital/Ruhr University Bochum, Herne
- Netherlands (5):
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Ziekenhuis St Jansdal, Harderwijk
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Twee Steden Ziekenhuis Vestiging Tilburg, Tilburg
- New Zealand (2):
  - Green Lane Hospital, Auckland
  - Wellington Cancer Centre, Wellington
- Spain (13):
  - Hospital de Cruces, Barakaldo, Bilbao
  - Hospital de la Santa Cruz I Sant Pau, Barcelona
  - Ciudad Sanitaria Vall D'Hebron, Barcelona
  - Hospital Clinic y Provincial de Barcelona, Barcelona
  - Hospital Nostra Senora Aranzazu, Donostia / San Sebastian
  - Hospital Universitario de Elche, Elche
  - Hospital de la Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario LA FE, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario Valencia, Valencia
  - Hospital Arnau Vilanova, Valencia
  - Hospital Miguel Servet, Zaragoza
- Switzerland (4):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Ratisches Kantons und Regionalspital, Chur
  - Kantonsspital - Saint Gallen, Sankt Gallen
- Royal Marsden Hospital, Sutton, England, United Kingdom

REFERENCES:
- [Result] Bottomley A, Debruyne C, Felip E, Millward M, Thiberville L, D'Addario G, Rome L, Zatloukal P, Coens C, Giaccone G. Symptom and quality of life results of an international randomised phase III study of adjuvant vaccination with Bec2/BCG in responding patients with limited disease small-cell lung cancer. Eur J Cancer. 2008 Oct;44(15):2178-84. doi: 10.1016/j.ejca.2008.06.036. PMID 18676140